CLINICAL TRIAL: NCT01007773
Title: Safety of Dexmedetomidine in Severe Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study will not be intiated
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Deborah Stein, Medical Director, Neurotrauma Critical Care; Chief, Section of Trauma Critical Care, R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HP-00042821; PRE-08-019
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Traumatic Brain Injury
Keywords: Dexmedetomidine; Intracranial Pressure; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dexmedetomidine; Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): In conjunction with conventional sedative and analgesic agents.
  Interventions: Drug: Precedex; Drug: Propofol
- Standard of Care (Active Comparator): Patients randomized to conventional sedation will have as the main pharmacologic agents to achieve sedation and analgesia propofol and fentanyl, respectively.
  Interventions: Drug: Propofol; Drug: Fentanyl

INTERVENTIONS:
Drug: Precedex — Once this patient is deemed stable on the propofol infusion, the patient will be started on a dexmedetomidine infusion at 0.4 mcg/kg/hr. The dexmedetomidine infusion will be titrated to a Richmond Agitation Sedation Scale (RASS) of 0 to -1 (maximum rate of 1.5 mcg/kg/hr). In the meantime, once sustained ICP control has been achieved, the initial sedative agent (usually propofol) will be weaned. Dexmedetomidine will be infused for up to 7 days or until removal of the ICP or when mechanical ventilation is discontinued. When the patient is ready to come off sedation, the dexmedetomidine will be weaned by 50% every hour over a 4-hour period to off.
  Other Names: Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Propofol — Propofol will be initiated at 25 mcg/kg/min and titrated to achieve an ICP < 20 mm Hg (up to a maximum of 75 mcg/kg/min). Propofol will be continued for up to 7 days or until removal of the ICP or when mechanical ventilation is discontinued.
  Other Names: Diprivan
  Arms: Standard of Care
Drug: Fentanyl — Fentanyl will be initiated and titrated to achieve adequate pain control.
  Other Names: Actiq; Fentora; Instanyl
  Arms: Standard of Care
Drug: Propofol — Propofol will be titrated to an ICP < 20 mm Hg until achievement of sustained ICP control.
  Other Names: Diprivan
  Arms: Dexmedetomidine

SUMMARY:
The aim of this study is to assess the safety and feasibility of dexmedetomidine as an adjunct to conventional sedative therapy compared to conventional sedative therapy alone in patients with severe traumatic brain injury.

DETAILED DESCRIPTION:
Approximately 52,000 deaths occur from traumatic brain injury (TBI) every year. TBI is a major cause of disability, death, and economic cost to our society. When the brain experiences injury, there is direct damage to the brain tissue causing local bleeding and bruising. This is called the primary injury. Additional damage, called secondary brain injury, can occur as a result of swelling of the brain, lack of oxygen to the brain, lowered blood pressure, and the release of inflammatory mediators. The type and degree of insults are major determinants in the final neurologic outcome of the patient who has sustained a TBI. Management of TBI is aimed at the prevention and treatment of these secondary insults.

The swelling of the brain following injury causes an increase in the pressure within the cranium. Increased pressure can reduce blood flow to parts of the brain, leading to further brain damage. An intracranial pressure (ICP) monitor measures the pressure surrounding the brain, and may be placed following traumatic brain injury to help evaluate swelling.

Agitation of the patient or exposure to painful stimuli may significantly increase ICP, and therefore, the use of sedative agents is important in ICP management. A variety of pharmacological agents have been suggested to treat agitation in the TBI patient. Unfortunately, no optimal sedative regimen has been identified for use in this patient population. One prospect is dexmedetomidine (Precedex®), which is FDA-approved for short-term (≤24 hours) sedation in the intensive care unit. Currently, to our knowledge, dexmedetomidine has not been studied prospectively in adults with traumatic brain injury. The safety and efficacy of dexmedetomidine are therefore unknown in severe TBI. Propofol is employed as a first-line sedative agent in neurotrauma patients due to its favorable pharmacokinetic profile. However, some patients require prolonged infusions and high rates of propofol. This has been shown increase their risk for development of a severe propofol-related infusion syndrome, which can be fatal.

Dexmedetomidine as an adjunct to existing conventional sedative therapy may help to facilitate decreasing the amount of other agents used, such as propofol. Therefore, the aim of this study is to assess the safety and feasibility of dexmedetomidine as an adjunct to conventional sedative therapy compared to conventional sedative therapy alone in patients with severe TBI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe traumatic brain injury, as defined by AIS score >2 for the head.
* Glasgow Coma Score (GCS) <9 on admission, or deterioration of GCS to <9 within 48 hours of admission due to traumatic brain injury.
* Placement of an intracranial pressure (ICP) monitor or intraventricular catheter (IVC) at the discretion of the Neurosurgical staff as part of standard of care.
* Patient is between 18 and 80 years of age, inclusive.

Exclusion Criteria:

* A body region, other than the brain, with an AIS score >2, or multiple system injury at the investigator's discretion.
* Glasgow Coma Score (GCS) >8 on admission or no decrease of GCS to <9 within 48 hours of admission.
* Placement of an ICP monitor or IVC not clinically indicated by Neurosurgical staff.
* Patient is under the age of 18, or over the age of 80.
* Determination of non-survivability due to the severity of brain injury.
* Non-English speaking, consentable LAR, or patient is non-English speaking.
* Patient is pregnant.
* Unable to obtain consent from a legally authorized representative (LAR).
* Patient is a prisoner, on parole or probation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial pressure | one week

SECONDARY OUTCOMES:
Doses of other sedatives | one week
Mortality | 6 months
GOS-E | 12 weeks, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Stein, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States